CLINICAL TRIAL: NCT02761707
Title: Biomarkers in Neural Disorders
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor
Other Study IDs: 827731
Record Dates: First submitted 2016-04-18; First posted 2016-05-04 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Parkinson's Disease; Alzheimer's Disease; Progressive Supranuclear Palsy; Essential Tremor; Multiple System Atrophy; Drug Induced Parkinson's Disease; Diffuse Lewy Body Disease; Myasthenia Gravis; Spinal Cord Injuries
MeSH Terms: conditions — Parkinson Disease; Alzheimer Disease; Supranuclear Palsy, Progressive; Essential Tremor; Multiple System Atrophy; Lewy Body Disease; Myasthenia Gravis; Spinal Cord Injuries | interventions — Neurofeedback

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (11):
- Parkinson's Disease: Non-smokers, ages 18-80, diagnosed with Parkinson's Disease. Must be Hoehn and Yahr stage 2 or less with a history of motor symptoms less than two years.
  Interventions: Other: Electrical Brainstem Responses; Other: Olfactory Tests; Other: Visual Deprivation; Other: Peripheral Nerve Stimulation
- Alzheimer's Disease: Non-smokers, ages 18-80, diagnosed with Alzheimer's Disease. Must meet the 2011 National Institute on Aging-Alzheimer's Association and the 1984 National Institute for Neurological and Communicative Disorders and Stroke-Alzheimer's disease and Related Disorders Association criteria for probable AD.
  Interventions: Other: Electrical Brainstem Responses; Other: Olfactory Tests; Other: Peripheral Nerve Stimulation
- Progressive Supranuclear Palsy: Non-smokers, ages 18-80, diagnosed with Progressive Supranuclear Palsy. Must meet the NINDS-SPSP criteria for probable PSP, which requires vertical supranuclear gaze palsy, prominent postural instability, and falls in the first year of onset, as well as a number of other clinical features.
  Interventions: Other: Electrical Brainstem Responses; Other: Olfactory Tests; Other: Peripheral Nerve Stimulation
- Essential Tremor: Non-smokers, ages 18-80, diagnosed with Essential Tremor.
  Interventions: Other: Electrical Brainstem Responses; Other: Olfactory Tests; Other: Peripheral Nerve Stimulation
- Drug-Induced Parkinson's Disease: Non-smokers, ages 18-80, diagnosed with Drug-Induced Parkinson's Disease.
  Interventions: Other: Electrical Brainstem Responses; Other: Olfactory Tests; Other: Peripheral Nerve Stimulation
- Myasthenia Gravis: Non-smokers, ages 18-80, diagnosed with Myasthenia Gravis.
  Interventions: Other: Electrical Brainstem Responses; Other: Olfactory Tests; Other: Peripheral Nerve Stimulation
- Multiple System Atrophy: Non-smokers, ages 18-80, who have been diagnosed with Multiple System Atrophy.
  Interventions: Other: Electrical Brainstem Responses; Other: Olfactory Tests; Other: Peripheral Nerve Stimulation
- Diffuse Lewy Body Disease: Non-smokers, ages 18-80, diagnosed with Diffuse Lewy Body Disease. Must meet the Consensus Criteria for the clinical diagnosis of DLBD.
  Interventions: Other: Electrical Brainstem Responses; Other: Olfactory Tests; Other: Peripheral Nerve Stimulation
- Healthy Controls: Non-smokers, ages 18-80, with no neurodegenerative disease, and no first-degree relatives with a neurodegenerative disease.
  Interventions: Other: Electrical Brainstem Responses; Other: Olfactory Tests; Other: Visual Deprivation; Other: Peripheral Nerve Stimulation
- Spinal Cord Injury
  Interventions: Other: Electrical Brainstem Responses; Other: Olfactory Tests; Other: Peripheral Nerve Stimulation
- Asymptomatic Relatives
  Interventions: Other: Electrical Brainstem Responses; Other: Olfactory Tests; Other: Peripheral Nerve Stimulation

INTERVENTIONS:
Other: Electrical Brainstem Responses — Eye blink responses will be induced using standard stimulating electrodes employed in surface electromyography (EMG). The subjects will recline with their eyes gently closed. Sticky electrodes will be placed to the left and below the left eye. 6 different facial regions will be stimulated. The electrical stimulation will be kept constant during the test sessions. To prevent habituation, the stimuli will be delivered randomly at intervals of 45-60 sec. Four 0.2 msec pulses will be presented. In some cases, paired pulse stimulation will be performed, and a conditioning stimulus will be applied to the target facial regions at the following intervals: 10, 200, 400, 600 and 800 msec. 4 pulses will be presented at each stimulus interval with randomized interval and pulse sequences.
  Other Names: Electromyography
Other: Olfactory Tests — Olfactory testing will be performed using standard tests. The University of Pennsylvania Smell Identification Test (UPSIT) assesses a subjects ability to identify odors in a forced choice format. The Snap and Sniff Threshold Test provides a threshold measure of phenyl ethyl alcohol. Short-term odor memory will be assessed using a standardized 12-item four-alternative forced-choice Odor Memory Test. This non-lexical test employs 10-, 30-, and 60-second delay intervals between the presentation of the target odorant and the first of four successively presented odors from which the target is to be selected.
Other: Visual Deprivation — During a 2-hour visual deprivation period, subjects will wear comfortable light-tight goggles with lenses that have been blackened by flat black paint. Subjects will be given the opportunity to recline comfortable in a padded reclining chair during this time.
  Groups: Healthy Controls; Parkinson's Disease
Other: Peripheral Nerve Stimulation — Electrical stimulation will be applied to a nerve of your arm. Sticky electrode pads will also be placed on a hand muscle. You will receive electrical stimulations that lasts less than a second. The stimulations will make your muscle twitch.
  Other Names: Repetitive Nerve Stimulation

SUMMARY:
This study seeks to establish the sensitivity and specificity of what appears to be a unique brainstem biomarker of Parkinson's Disease (PD) - an electrically induced olygosynaptic nasotrigeminal reflex response - in differentiating early stage PD from normal controls and from patients with various other neurodegenerative diseases. This study will additionally compare the biomarker to olfactory testing.

DETAILED DESCRIPTION:
Parkinson's disease (PD), a devastating age-related disease that is clinically defined by its effects on the motor system, afflicts more than six million people worldwide, imposing enormous burdens on patients, relatives, caretakers, and society in general. Diagnostic errors are common, particularly as symptoms first arise. The most common misdiagnoses are Alzheimer's disease (AD), essential tremor, and vascular pseudo-Parkinson's Disease. An accurate diagnosis is typically made at a later stage of the disease when marked and irreversible damage has occurred within the motor control system of the brain. Sensitive and specific biomarkers of the early stages of PD are urgently needed. Identification of such markers is critical for the development and assessment of medications and other interventions designed to eliminate or reduce the gradual and irreversible decline of neurons involved in the disorder. This study seeks to establish the sensitivity and specificity of what appears to be a unique brainstem biomarker of PD - an electrically induced trigeminal nerve blink reflex response - in differentiation of early stage PD from normal controls and such neurodegenerative diseases as early stage AD, progressive supranuclear palsy (PSP), and diffuse Lewy Body disease (DLBD). This study will additionally compare the biomarker to olfactory test results.

ELIGIBILITY:
Inclusion Criteria:

* The Parkinson's disease (PD) patients will be Hoehn and Yahr stage 2 or less with a history of motor symptoms less than two years.
* The Alzheimer's disease (AD) patients will meet the 2011 National Institute on Aging-Alzheimer's Association and the 1984 National Institute for Neurological and Communicative Disorders and Stroke-Alzheimer's disease and Related Disorders Association criteria for probable AD.
* The progressive supranuclear palsy (PSP) patients will have met the NINDS-SPSP criteria for probable PSP, which requires vertical supranuclear gaze palsy, prominent postural instability, and falls in the first year of onset, as well as a number of other clinical features.
* The DLBD patients will meet the Consensus Criteria for the clinical diagnosis of DLBD.
* The healthy controls will be matched to the PD patients on such variables as sex, age, education level, and ethnicity.
* The essential tremor (ET), multiple system atrophy (MSA), myasthenia gravis (MG), multiple system atrophy (MSA), Parkinson's disease dementia (D-PD), and Spinal Cord Injury (SCI) patients will meet the generally-accepted diagnostic criteria for these disorders.

Exclusion Criteria:

* Drug abuse.
* Any other known and potentially confounding condition that could reasonably be expected to interfere with the study assessments.
* Under age 18.
* Over age 80.
* Smoker.
* Pregnant or nursing.
* Healthy control with a first degree relative who has a neurodegenerative disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal controls and patients with such neural disorders as Parkinson's Disease(PD), Alzheimer's disease (AD), progressive supranuclear palsy (PSP), essential tremor (ET), dementia with Parkinson's disease (D-PD), myasthenia gravis (MG), multiple system atrophy (MSA), diffuse Lewy body disease (DLBD), and Spinal Cord Injury (SCI). None will be cigarette smokers. The patients will be diagnosed accord to current consensus criteria. The healthy controls will be matched to the PD patients on such variables as sex, age, education level, and ethnicity. The Healthy Controls will be asked to answer questions regarding the disease state of their first degree family members to ensure that these first degree family members do not have a neurodegenerative diseases. Every effort will be made to include women and minority subjects.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
Latency, amplitude, and area under the curve of brainstem reflex response | 1 Hour
  Latency, amplitude, and area under the curve of electrical brainstem reflex response of trigeminal nerve branches measured on the face musculature (before and after short-term visual deprivation).
Score on the University of Pennsylvania Smell Identification Test | 20 Minutes
  The number of correct odor identification responses out of 40 from the standardized University of Pennsylvania Smell Identification Test (before and after short-term visual deprivation).
Score on the Odor Discrimination/Memory Test | 30 Minutes
  The number of correct responses in picking out an odor previously presented from three foils 10, 30, and 60 sec later using the standardized Odor Detection/Discrimination Test (before and after short-term visual deprivation).
Score on an Odor Detection Threshold Test | 20 Minutes
  The average of 7 reversals in a staircase odor detection threshold test that employs phenyl ethyl alcohol (rose oil) concentrations ranging from -7 to -2 log dilutions in light mineral oil.

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Doty, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No